CLINICAL TRIAL: NCT05443776
Title: In Vivo Investigation of Six Different Membranes Including Their Physical, Chemical and Biological Properties - a Pilot Study.
Brief Title: In Vivo Investigation of 6 Membranes Including Their Physical, Chemical and Biological Properties.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Jordi caballé, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: CIR-ECL-2018-03
Record Dates: First submitted 2022-03-18; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Bone Regeneration; Tissue Engineering

STUDY DESIGN:
Intervention Model Description: 6 different. products used, each compared between each other
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Study group biomaterial 1 (Experimental)
  Interventions: Other: Biomaterial implantation
- Study group biomaterial 2 (Experimental)
  Interventions: Other: Biomaterial implantation
- Study group biomaterial 3 (Experimental)
  Interventions: Other: Biomaterial implantation
- Study group biomaterial 4 (Experimental)
  Interventions: Other: Biomaterial implantation
- Study group biomaterial 5 (Experimental)
  Interventions: Other: Biomaterial implantation
- Study group biomaterial 6 (Experimental)
  Interventions: Other: Biomaterial implantation

INTERVENTIONS:
Other: Biomaterial implantation — Implant a approved biomaterial by European Regulatory Agencies

SUMMARY:
A wide range of resorbable and non-resorbable membranes have been investigated over the last decades. Barrier membranes protect bone defects from ingrowth of soft tissue cells, provide mechanical stability of the defect area and allow bone progenitor cells to develop within a blood clot that is formed beneath the barrier membrane, taking a minimum of four to six weeks for periodontal tissues and 16-24 weeks for bone1,2.These membranes are utilized to reconstruct bone defects prior to implantation and to cover dehiscences and fenestrations around dental implants.

When aiming to regenerate bone, resorbable or a non - resorbable membranes should be selected depending on location, size and defect area. However, until now the ideal membrane has not been described due to different opinions between authors3,4. Nevertheless, an ideal membrane should maintain its barrier function enough time for new bone formation, and if possible should be resorbable, so that a second surgical procedure for the explantation of the membrane would not be required, thus reducing the morbidity5. However, the use of a barrier membrane is a technique-sensitive procedure that is not free of complications. The main cause of Guided Bone Regeneration (GBR) failure is related to early or late exposure of the membrane, leading to contamination and infection of the biomaterial, irreversibly compromising bone regeneration4,6,7. Consequently, the inflammatory reaction of the surrounding soft tissues may require early removal of the membrane. Other complications, such as the onset of an abscess with purulent exudate, can also lead to a complete failure of GBR even without exposure of the membrane.

It is thought necessary to perform this clinical study due to the lack of information present in the literature about the different types of membranes that exist nowadays, how they act in the human body with or without performing some type of regeneration and how our body acts towards them.

ELIGIBILITY:
* Inclusion Criteria:
* Overall, healthy patients that qualify for oral surgery (ASA I and II)
* Older than 18 years old
* Requiring extraction of 1-3 teeth (premolars or molars) that do not involve the aesthetic area
* Stable post-extraction socket walls with at least 4 walls
* Patient candidate to an early implant placement in the extraction area
* Informed consent signed
* Adequate oral hygiene: plaque index < 25% before the surgery
* Smoker of <10 cigarettes per day
* Able to follow the instructions and able to meet the follow-ups
* Healthy or controlled periodontal disease
* Exclusion Criteria:
* Patients who not agree with informed consent
* Untreated periodontal disease
* Presence of dehiscence and/or fenestration at buccal plate of the extraction teeth
* Patient who will need GBR or Block Regeneration
* after the extraction
* History of head and/or neck radiation
* History of chemotherapy in the five years prior of the surgery
* Non controlled Diabetes
* Chronic corticoids or other medication that may influence healing and / or osseointegration
* Smoker of >10 cigars per day
* Alcohol or other drugs abuse
* Patient going under bisphosphonates treatment or taking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Grade of the biocompatibility of the biomaterials | Outcome will be measured once, after samples are collected and processed, 2-3 months after implantation.
  The grade of biocompatibility will be assessed by using histology tools, analyzing the type of cells present in the sample.
Characteristics of the inmune response of the biomaterials in the host tissues | Outcome will be measured once, after samples are collected and processed, 2-3 months after implantation.
  The characteristics of the inmune response will be assessed by using histology tools, determining the presence of inflammatory cells such as macrophages.
Rate of degradation of the biomaterials | Outcome will be measured once, after samples are collected and processed, 2-3 months after implantation.
  The rate of degradation of the biomaterials will be assessed by using histology tools, analyzing the amount of biomaterial present in the samples and comparing it to the amount that was implanted.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Caball, DDS MSc PhD, Principal Investigator — UIC Barcelona
Locations (1):
- UIC Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No